CLINICAL TRIAL: NCT06300047
Title: Aiming for Something Sweeter: Supporting Youth With Type 1 Diabetes During Transition From Pediatric to Adult Diabetes Care
Brief Title: Diabetes Transition Coordinator Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: REB23-0679
Record Dates: First submitted 2023-11-01; First posted 2024-03-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The usual care group is defined as the group who receives usual care and serves as the control group. This group is defined prior to the implementation of the intervention. We include a two month wash out period between our two groups to avoid care providers 'holding on' to patients they feel may benefit from the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (No Intervention): No intervention group used as a control leading into the intervention for comparative analysis. Patients in this arm receive care as usual with no changes and are not aware of the intervention group.
- Intervention Group (Experimental): Patients in this arm receive access to and support from a Transition coordinator who will meet with them prior to transition from pediatric to adult care and follow up with them every 2 months throughout the first year of their transition period utilizing phone, text, email, social media.
  Interventions: Other: Non-Medical Transition Coordinator

INTERVENTIONS:
Other: Non-Medical Transition Coordinator — Participants in this intervention arm will have access to the non-medical transition coordinator to support their transition from pediatric to adult care.
  Arms: Intervention Group

SUMMARY:
The goal of this interventional study is to assess the effects and evaluate the implementation of a pediatric to adult care transition intervention in youth with T1D on clinical, patient-reported, and implementation outcomes, including an economic analysis.

The 3 main aims are:

1. To assess the effects of our transition intervention on clinical and patient-reported outcomes.
2. To implement the transition intervention and evaluate the implementation outcomes.
3. To evaluate the economic impacts of the transition intervention. Participants will have access to a transition coordinator before, during, and after their planned transition from pediatric to adult care as standard of care.

Researchers will compare a pre-intervention cohort to evaluate the impact of the transition coordinator intervention.

DETAILED DESCRIPTION:
Both usual care and intervention groups will receive routine diabetes care as per Canadian national guidelines. Usual care (routine care) includes regular appointments with their pediatric diabetes care team (i.e., pediatric endocrinologist, diabetes nurse or dietician) and post-transfer with their adult diabetes team (i.e., physician and as needed visits with a diabetes educator and/or a dietician). The transition process usually starts at age 14 with discussions during clinic with youth and families around increased autonomy, self-care, organization of adult healthcare services and specific transition topics such as driving, drugs, alcohol, relationships, finances and living away from home.

The usual care group is defined as the group who receives usual care and serves as the control group. This group is defined prior to the implementation of the intervention. We include a two month wash out period between our two groups to avoid care providers 'holding on' to patients they feel may benefit from the intervention.

The intervention group (in addition to usual care) is provided additional support by way of a non-medical transition coordinator during the transition and transfer from pediatric to adult diabetes care. The non-medical transition coordinator encourages problem solving, self-management skills, and supports navigating the 'adult world'. In the year prior to transfer, the transition coordinator will meet each participant in person or virtually once during their routine pediatric diabetes appointment to explain their role prior to transfer. The transition coordinator role includes the following tasks: (1) use of text messaging, email, or phone communication (as per participant's preference) to maintain contact with the participant every 2 months for 12 months past the transfer date; (2) use of text messaging, email, or telephone as needed when participants reach out to them to answer any questions whereby the transition coordinator would provide direction; (3) assisting participants with finding family physicians (if needed); (4) assisting with completion of financial assistance, disability, insurance forms; (4) addressing any stated psychosocial needs by relaying information on community supports for participants and families; and, (5) maintaining a private Facebook® page and a transition website in which participants were encouraged to use. Website contents include information on transition, adult diabetes care (i.e., location, contact numbers, what to expect in adult care), diabetes resources as well as mental health resources. The website will be updated to have information relevant to each implementation site. We may add other types of social media to share information about transition (i.e., TikTok, Instagram), and this will be considered during our pre-implementation phase. The transition coordinator will not provide any medical advice or counselling.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of T1D according to Diabetes Canada's guidelines for at least 12 months
* aged 17 to 18 years
* have had an appointment with their pediatric endocrinologist in the last 12 months
* in the last year of pediatric care and transferring to adult care in Alberta within the next year
* English proficiency (for surveys)
* Personal Health Number (PHN) for data linkage.

Exclusion Criteria:

-

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Lost to Followup | within 1 year of transfer date from pediatric care
  % of participants who are lost to follow up as defined by not attending at least one routine clinic visit in adult diabetes care with a health care professional to be ascertained from physician billing claims or NACRS claims data

SECONDARY OUTCOMES:
Patient Reported Outcome Survey 1 | within 2 months of transfer from pediatric care, repeated at 12 months after transfer
  Problem Areas in Diabetes - Teen version Survey
Patient Reported Outcome Survey 2 | within 2 months of transfer from pediatric care, repeated at 12 months after transfer
  Diabetes Self-Efficacy Survey
Patient Reported Outcome Survey 3 | within 2 months of transfer from pediatric care, repeated at 12 months after transfer
  Diabetes Quality of Life for Youth Survey (short version)
Clinical Outcome 1 | one year prior to transfer from pediatric care up to 18 months post transfer
  mean total number of clinic visits with any health care professional collected from NACRS claims data and physician claims data
Clinical Outcome 2 | one year prior to transfer from pediatric care up to 18 months post transfer
  total number of diabetes related emergency department visits and hospitalizations for diabetic ketoacidosis
Clinical outcome 3 | one year prior to transfer from pediatric care up to 18 months post transfer
  mean HbA1c
Clinical outcome 4 | one year prior to transfer from pediatric care up to 18 months post transfer
  total number of HbA1c tests completed
Clinical Outcome 5 | one year prior to transfer from pediatric care up to 18 months post transfer
  mean urinary albumin:creatinine ratio
Clinical Outcome 6 | one year prior to transfer from pediatric care up to 18 months post transfer
  total number of urinary albumin:creatinine ratio tests completed

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Butalia, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No